CLINICAL TRIAL: NCT02452827
Title: The Correlation of Myodural Bridges to Biomechanical Parameters in Patients Suffering From Primary Chronic Neck Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0034-15
Record Dates: First submitted 2015-05-18; First posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Primary Chronic Neck Pain: Patients suffering for at least 3 years from neck pain without any underlying pathology who have undergone MRI. Biomechanical parameters of neck movements will be investigated.
  Interventions: Other: Biomechanical parameters; Other: MRI
- Control: Patients without neck pain who have undergone MRI for any reason. Biomechanical parameters of neck movements will be investigated.
  Interventions: Other: Biomechanical parameters; Other: MRI

INTERVENTIONS:
Other: Biomechanical parameters
Other: MRI — MRI of cervical spine

SUMMARY:
In recent years, an anatomical connection of suboccipital muscle fibers to the dura has been found in pathological studies. The physiologic function of these fibers is still unknown. Using Magnetic Resonance Tomography (MRI), this study will investigate whether these fibers undergo changes in patients suffering from primary chronic neck pain. In addition, the biomechanical parameters of neck movements in these patients will be correlated with the imaging findings.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Neck Pain

Exclusion Criteria:

* Have undergone cervical spine surgery
* Known cerebral vascular disease of the carotid or vertebral arteries
* Malignant disease of the cervical spine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Primary Chronic Neck Pain who have undergone MRI. Healthy volunteers who have undergone MRI of the cervical spine.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Volume and Number of Muscle Fibers in Myodural Bridges | One hour
  A composite outcome including the interpretation, counting and measurement of muscle fibers as found on MRI

SECONDARY OUTCOMES:
Measurement of cervical range of motion | Two hours
  Measurements will be made using a cervical range of motion device (CROM Device)

CONTACTS AND LOCATIONS:
Overall Officials: Yaron River, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel